CLINICAL TRIAL: NCT03981172
Title: Effects of Daily Snack Food Intake on Food Reinforcement Depend on Weight Status and Energy Density
Brief Title: Food Reinforcement, Weight Status, and Energy Density
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jennifer Temple, Associate Professor, State University of New York at Buffalo
Other Study IDs: Temple10132009
Record Dates: First submitted 2011-03-24; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Reinforcing Value of Food
Keywords: food reinforcement; food liking; motivation; dopamine; obesity; energy density; snacks
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Non-obese/HED: Non-obese women given 60 gram portions of high energy density snack foods to consume daily for two weeks.
  Interventions: Behavioral: Daily snack food intake
- Non-Obese/LED: Non-obese participants that were given 60 gram portions of low energy density foods to consume daily for two weeks.
  Interventions: Behavioral: Daily snack food intake
- Obese/LED: Obese participants that were given 60 gram portions of low energy density snack foods to consume daily for two weeks.
  Interventions: Behavioral: Daily snack food intake
- Obese/HED: Obese participants that were given 60 gram portions of high energy density snack foods to consume daily for two weeks.
  Interventions: Behavioral: Daily snack food intake

INTERVENTIONS:
Behavioral: Daily snack food intake — participants consumed 60 gram portions of either low energy density or high energy density snack foods every day for two weeks.

SUMMARY:
The investigators previous studies have shown that obese and non-obese individuals respond differently to daily intake of snack food. The purpose of this study was to determine whether these differences are specific to high energy density snack foods. The investigators hypothesized that obese individuals would show an increase in motivation to obtain high energy density snack foods after two weeks of daily consumption, but that non-obese women and obese women consuming low energy density foods would have reduced motivation to consume snack foods after two weeks of daily consumption.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 50 years old, female, like study foods.

Exclusion Criteria:

* current smoker, currently on a diet, medical conditions or medication affecting appetite (ex. methylphenidate).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women ages 18 - 50 were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Number of operant responses | about one month
  Participants were asked to click a mouse button to gain access to food. A point was earned after a certain number of button presses and after 5 points were earned, the participant received 100 kcal portion of food.

SECONDARY OUTCOMES:
Food liking | about one month
  participants rated how much they liked the food on a Likert-type scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States